CLINICAL TRIAL: NCT02934685
Title: A Phase III Randomized Study of Hypofractionated Image-guided Volumetric Modulated Arc Radiotherapy (IG-VMAT) Versus Conventionally Fractionated IG-VMAT in Patients With Localized Prostate Cancer
Brief Title: IG-VMAT for Localized Prostate Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Gaofing Li, director of radiotherapy department, Beijing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BeijingH-01-RT
Record Dates: First submitted 2016-07-11; First posted 2016-10-17 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Prostate Cancer
Keywords: Prostatic Neoplasms; radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hypofraction (Experimental): 70 Gy in 28 fractions over 5.6 weeks
  Interventions: Radiation: hypofraction
- convention (Active Comparator): 80Gy in 40 fractions over 8 weeks
  Interventions: Radiation: convention

INTERVENTIONS:
Radiation: hypofraction — 70 Gy in 28 fractions over 5.6 weeks
  Arms: hypofraction
Radiation: convention — 80Gy in 40 fractions over 8 weeks
  Arms: convention

SUMMARY:
To determine if hypofractionated IG-VMAT (70 Gy in 28 fractions over 5.6 weeks) will result in disease-free survival (DFS) that is no worse than DFS following conventionally fractionated IG-VMAT (80Gy in 40 fractions over 8 weeks) in patients treated for localized prostate cancer. Analysis the local progression, disease-specific survival (DFS), freedom from biochemical recurrence (FFBR), and overall survival (OS) of two groups. Observe the incidence of GI and GU toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-79
* Histologically confirmed prostate adenocarcinoma
* Clinical stage T1-3N0M0 according to the AJCC 6th edition
* Gleason score must be >5
* KPS >70
* No radical surgery or cryosurgery for prostate cancer

Exclusion Criteria:

* Prior or concurrent invasive malignancy (except non-melanomatous skin cancer) or lymphomatous/hematogenous malignancy unless continually disease free for a minimum of 5 years. (For example, carcinoma in situ of the bladder or oral cavity is permissible)
* Evidence of distant metastases
* Previous radical surgery (prostatectomy) or cryosurgery for prostate cancer
* Previous pelvic irradiation, prostate brachytherapy, or bilateral orchiectomy
* Previous or concurrent cytotoxic chemotherapy for prostate cancer

Ages: 50 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-02 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Biochemical progression free survival | up to 18 months
  Number of participants who are free of biochemical relapse after a specified duration of time.Phoenix definition of biochemical failure.

SECONDARY OUTCOMES:
Incidence of "acute" adverse events as assessed by NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v. 4.0 | From the start of radiation therapy (RT) to first occurrence of worse severity of adverse event within 30 days after the completion of RT
Time to "late" grade 2+ adverse events as assessed by NCI CTCAE v. 4.0 | From the date of completion of RT to the date of first grade 2 or above adverse event occurring 30 days after the completion of RT
Overall Survival | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Gaofeng Li, director, Principal Investigator — Beijing Hospital
Locations (1):
- Beijing Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No